CLINICAL TRIAL: NCT00026208
Title: Risk-Adapted Stanford V-C With Radiotherapy for Clinical Stage I and IIA Favorable Hodgkin's Disease: The G5 Study
Brief Title: Combination Chemotherapy Plus Low-Dose Radiation Therapy in Treating Patients With Stage I or Stage IIA Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ranjana Advani, Saul A. Rosenberg, MD, Professor of Lymphoma, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13081; LYMHD0002 (Other: OnCore)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Lymphoma, Hodgkin Disease; Lymphoma; Hodgkin Disease; Lymphoma: Hodgkin
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Vincristine; Vinblastine; Cyclophosphamide; Doxorubicin; Prednisone; Bleomycin; Etoposide; etoposide phosphate; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Patients with tumors 5 to 10 cm were to be assigned to concurrent radiotherapy, and participants with tumors less than 5 cm were initially planned to not receive radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stanford V-C + Low-dose Radiotherapy (Experimental): "Sanford V-C" = Vinblastine, cyclophosphamide, doxorubicin, prednisone, bleomycin, + etoposide.
  Radiotherapy = 20 Gy modified involved field radiotherapy
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Bleomycin; Drug: Etoposide; Radiation: Low-dose radiotherapy (RT)
- Stanford V-C only (Experimental): "Sanford V-C" = Vinblastine, cyclophosphamide, doxorubicin, prednisone, bleomycin, + etoposide.
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Bleomycin; Drug: Etoposide

INTERVENTIONS:
Drug: Vincristine — 1.4 mg/m² intravenously (IV) on week 2, 4, 6, 8
  Other Names: Vinblastine; Leurocristine sulfate; Oncovin; Vincasar; LCR; VCR; Vincristin; Vincristina; Vincristinum; 22-Oxovincaleukoblastin; 22-Oxovincaleukoblastine
Drug: Cyclophosphamide — 650 mg/m², on week 1 and 5
  Other Names: Cytoxan; Neosar; Cyclophosphamidum; Cyclophosphamid; Ciclofosfamida; Cytophosphane; Ledoxina; Bis(2-chloroethyl)phosphoramide cyclic propanolamide ester; 2-[Bis(2-chloroethylamino)]-tetrahydro-2H-1,3,2-oxazaphosphorine-2-oxide; N,N-Bis(2-chloroethyl)tetrahydro-2H-1,3,2-oxazaphosphorin-2-amine 2-oxide
Drug: Doxorubicin — 25 mg/m², on week 1, 3, 5, 7
  Other Names: Adriamycin; Doxorubicinum; Doxorubicine; Rubex; Hydroxydaunomycin HCl; Hydroxydoxorubicin HCl; Hydroxydaunorubicin; 14-hydroxydaunomycin; 14-hydroxydaunorubicine; (1S,3S)-3-Glycoloyl-3,5,12-trihydroxy-10-methoxy-6,11-dioxo-1,2,3,4,6,11-hexahydrotetracen-1-yl 3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranoside; (8S-cis)-10-((3-amino-2,3,6-Trideoxy-alpha-L-lyxo-hexopyranosyl)oxy)-7,8,9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-5,12-naphthacenedione
Drug: Prednisone — 40 mg/m², oral, every other day. Taper-reduction 10 mg/m² every other day during last 2 weeks of chemotherapy
  Other Names: Dehydrocortisone; Deltasone; Liquid Pred; Meticorten; Orasone; Prednicot; predniSONE Intensol; Rayos; Sterapred; Prednisona; Prednisonum; 1,2-Dehydrocortisone; 1,4-Pregnadiene-17alpha,21-diol-3,11,20-trione; 17,21-Dihydroxypregna-1,4-diene-3,11,20-trione
Drug: Bleomycin — 5 u/m² intravenously (IV) on week 2, 4, 6, 8
  Other Names: Bleomycin A2; Bleomycine; Bleocin; Bleomicin; Bleomicina; Bleomycinum; BLM
Drug: Etoposide — 60 mg/m² x 2 intravenously (IV) on week 3, 7 (d 15, 16, 43, 44)
  Other Names: Toposar; Etopophos; Vepesid; VP-16; Etoposido; Etoposidum; trans-Etoposide; 4-demethylepipodophyllotoxin β-D-ethylideneglucoside; 4'-Demethylepipodophyllotoxin 9-(4,6-O-(R)-ethylidene-beta-D-glucopyranoside); 9-((4,6-O-Ethylidine-beta-D-glucopyranosyl)oxy)-5,8,8a,9-tetrahydro-5-(4-hydroxy-3,4-dimethyloxyphenyl)furo(3',4'':6,7)naptho-(2,3-d)-1,3-dioxol-6(5aH)-one
Radiation: Low-dose radiotherapy (RT) — 20 Grey (Gy) modified involved field radiotherapy administered as consolidative irradiation will beginning between 2 and 12 weeks after the completion of Stanford V-C chemotherapy regimen.
  Arms: Stanford V-C + Low-dose Radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: This phase 2 trial is studying how well giving combination chemotherapy together with low-dose radiation therapy works in treating patients with stage I or stage IIA Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the freedom from progression in patients with stage I or IIA Hodgkin's lymphoma with a favorable prognosis treated with "Stanford V-C" chemotherapy comprising cyclophosphamide, doxorubicin, vinblastine, prednisone, vincristine, bleomycin, and etoposide with low-dose radiotherapy (RT).
* Minimize the early and late effects of treatment in these patients by avoiding staging laparotomy and its consequences, limiting cumulative doses of chemotherapy, and reducing the dose of RT to moderately bulky sites of disease.
* Assess early and late treatment-related toxicity, freedom from second disease progression, and overall survival at 5 and 10 years in patients treated with this regimen.

Participants receive Stanford V-C chemotherapy comprising cyclophosphamide IV over 30 to 60 minutes weekly on weeks 1 and 5; doxorubicin IV and vinblastine IV over 5 minutes once weekly on weeks 1, 3, 5, and 7; oral prednisone every other day on weeks 1 to 8; vincristine IV, and bleomycin IV over 5 minutes once weekly on weeks 2, 4, 6, and 8; and etoposide IV over 60 minutes on days 1 and 2 of weeks 3 and 7. Prior to protocol amendment, participants were assigned to treatment on the basis of tumor size (< 5 cm vs 5 to 10 cm), with only the participants with larger tumors receiving RT. Beginning 2 to 3 weeks after completion of chemotherapy, participants in the +RT group will receive low-dose radiotherapy 5 days a week for approximately 3 weeks. Subsequent to amendment, all participants received RT.

Participants are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of previously untreated stage I or IIA Hodgkin's lymphoma, eligible subtypes

  * Nodular sclerosis
  * Mixed cellularity
  * Classical, not otherwise specified
* Age ≥ 18 years and ≤ 70 years
* Granulocytes ≥ 2 x 10e6/µL
* Platelets ≥ 150 x 10e6/µL
* Bilirubin ≤ 2.5 mg/dL
* Serum creatinine ≤ 2 mg/dL
* Patients > 50 years or those with a history of cardiac disease should have an ejection fraction ≥ 50%
* All scans, X-rays, laboratory tests must be performed within 6 weeks of enrollment
* Pathologic material reviewed at Stanford University
* Evaluation by Stanford Medical Oncology and Radiation Oncology with review at the Hodgkin's Disease Staging Conference
* Written informed consent

EXCLUSION CRITERIA:

* Lymphocytic predominance Hodgkin's disease
* Prior treatment for Hodgkin's disease
* Mediastinal mass equal to or greater than one-third the maximum intrathoracic diameter on a standing posteroanterior chest x-ray
* Any lymph node mass > 10 cm in greatest trans-axial diameter
* Two or more extranodal sites of disease
* Constitutional (B) symptoms present at diagnosis
* Prior or concurrent malignancies within 5 years (EXCEPTION: basal cell carcinoma of the skin)
* Any medical contraindication to the planned treatment, including:

  * Pregnant
  * Positive antibody test for the human immunodeficiency virus (HIV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2001-06; Primary Completion 2013-04-26 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjana H Advani, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Kaiser Permanente Medical Center, Vallejo, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stanford V-C + Low-dose Radiotherapy: "Stanford V-C" = Vinblastine, cyclophosphamide, doxorubicin, prednisone, bleomycin, + etoposide.
  * Vincristine: 1.4 mg/m² intravenously (IV) on week 2, 4, 6, 8
  * Cyclophosphamide: 650 mg/m², on week 1 and 5
  * Doxorubicin: 25 mg/m², on week 1, 3, 5, 7
  * Prednisone: 40 mg/m², oral, every other day. Taper-reduction 10 mg/m² mg every other day during last 2 weeks of chemotherapy
  * Bleomycin: 5 u/m² intravenously (IV) on week 2, 4, 6, 8
  * Etoposide: 60 mg/m² x 2 intravenously (IV) on week 3, 7 (d 15, 16, 43, 44)
  "Low-dose radiotherapy (RT)" = 20 Grey (Gy) modified involved field radiotherapy administered as consolidative irradiation will beginning between 2 and 12 weeks after the completion of Stanford V-C chemotherapy regimen.
- Stanford V-C Only: "Stanford V-C" = Vinblastine, cyclophosphamide, doxorubicin, prednisone, bleomycin, + etoposide.
  * Vincristine: 1.4 mg/m² intravenously (IV) on week 2, 4, 6, 8
  * Cyclophosphamide: 650 mg/m², on week 1 and 5
  * Doxorubicin: 25 mg/m², on week 1, 3, 5, 7
  * Prednisone: 40 mg/m², oral, every other day. Taper-reduction 10 mg/m² mg every other day during last 2 weeks of chemotherapy
  * Bleomycin: 5 u/m² intravenously (IV) on week 2, 4, 6, 8
  * Etoposide: 60 mg/m² x 2 intravenously (IV) on week 3, 7 (d 15, 16, 43, 44)
Period: Overall Study
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Started | 72 | 4
Completed | 71 | 4
Not Completed | 1 | 0
Not completed — Complications of auto accident | 1 | 0

BASELINE CHARACTERISTICS:
Population: Prior to amendment, participants with tumor size < 5 cm received Stanford V-C only. Subsequent to amendment, all participants received Stanford V-C + low-dose radiotherapy (RT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only | Total
Number analyzed (Participants) | 72 | 4 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 4 | 74
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 2 | 45
  Male | 29 | 2 | 31
Region of Enrollment [Number; unit: participants]
  United States | 72 | 4 | 76

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was assessed for 3 years from the completion of treatment. Progression-free survival was considered to mean the proportion of patients (percentage) still alive without disease recurrence or progression.
Time Frame: up to 3 years
Population: Does not include those participants whose treatment was significantly modified due to accidental injury; or who were lost-to-follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 70 | 4
percentage of participants | 89.7 | 50

2. Secondary Outcome: Frequency of Complete Response
Description: The frequency of complete response (CR) is reported as the number (proportion) of subjects in complete response, as assessed during weeks 4 to 5 of chemotherapy. Per protocol, CR is defined as "complete regression of all palpable and radiographic demonstrable disease" by computed tomography (CT) scan or positron emission tomography-CT (PET-CT).
Time Frame: 5 weeks
Population: Participants, for whom a PET-CT scan was not conducted in week 4 to 5 of treatment, were not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 38 | 0
Participants | 31 |

3. Secondary Outcome: Early Treatment-related Toxicity
Description: Early treatment-related toxicity was assessed as the number of treatment-related, non-serious adverse events that occurred during treatment or within 30 days of the completion of treatment.
Time Frame: Within 30 days of treatment
Measure: Number; unit: treatment-related adverse events
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 72 | 4
treatment-related adverse events | 422 | 24

4. Secondary Outcome: Late Treatment-related Toxicity
Description: Late treatment-related toxicity was assessed as the overall number of late-appearing toxicities (ie, related adverse events, after treatment completion) including but not limited to diagnosis of a 2nd cancer; hypothyroidism; infertility; pulmonary toxicity; or cardiac toxicity, at up to 16 years from date of diagnosis.
Time Frame: 16 years
Measure: Number; unit: treatment-related adverse events
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 72 | 4
treatment-related adverse events
  Second Cancer | 2 | 0
  Hypothyroidism | 19 | 0

5. Secondary Outcome: Second Hodgkin's Disease Progression
Description: Second Hodgkin's disease progression is reported as the number of participants experiencing 2 instances of progression of the underlying Hodgkin's disease, assessed at up to 16 years from date of diagnosis.
Time Frame: 16 years
Population: Data to confirm Hodgkin's disease 2nd progression was not available for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 69 | 4
Participants | 3 | 1

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was assessed at up to 16 years from date of diagnosis, and reported as the median years of survival with standard deviation.
Time Frame: 16 years
Population: Includes all participants, except those whose treatment was significantly modified due to accidental injury. Subjects who became lost-to-follow-up were censored at their last known value.
Measure: Median (Full Range); unit: years
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 71 | 4
years | 10.4 [0.7 to 15.5] | 13.2 [1.8 to 13.9]

7. Secondary Outcome: Survival at 5 and 10 Years
Description: Survival at 5 and 10 years is expressed at the percentage of subjects known to remain alive at those timepoints.
Time Frame: 5 and 10 years
Population: For overall survival at 5 and 10 years, this analysis does not include those participants known to be alive, but whose diagnosis was less than 5 or 10 years prior to current date or last date known alive, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
Number analyzed (Participants) | 69 | 4
Participants
  5 years | 67 | 3
  10 years: number analyzed (Participants) | 46 | 4
  10 years | 41 | 3

ADVERSE EVENTS:
Time Frame: 16 years
Arm/Group | Stanford V-C + Low-dose Radiotherapy | Stanford V-C Only
All-Cause Mortality (participants affected / at risk) | 7/72 | 0/4
Serious Adverse Events (participants affected / at risk) | 25/72 | 2/4
Other Adverse Events (participants affected / at risk) | 72/72 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanford V-C + Low-dose Radiotherapy (N=72) | Stanford V-C Only (N=4)
Hypothyroidism (Endocrine disorders) | 17 (17) | 2 (2)
Second cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Crush injury, automobile accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fever (General disorders) | 5 (6) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanford V-C + Low-dose Radiotherapy (N=72) | Stanford V-C Only (N=4)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Secondary to automobile accident
Lymphocyte count decreased (Investigations) | 55 (101) | 4 (11)
Fatigue/Malaise (General disorders) | 58 (58) | 3 (3)
Fever (General disorders) | 3 (3) | 0 (0)
Nausea and Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Metallic Taste in Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection with grade 3 ANC grade 2 ATT (no hospitalization) (Blood and lymphatic system disorders) | 1 (1) | 0
Oral Mucositis (Gastrointestinal disorders) | 7 (7) | 0 (0)
Mild Oral Sensitivity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Toxicity (Gastrointestinal disorders) | 8 (8) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 26 (26) | 1 (1)
Acute Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 27 (27) | 0 (0)
Tenderness at the PICC site (General disorders) | 1 (1) | 0 (0)
Discomfort, burning & increased sensitivity (General disorders) | 1 (1) | 0 (0)
PICC line removed (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 51 (51) | 2 (2)
Constipation (Gastrointestinal disorders) | 40 (40) | 3 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 40 (40) | 3 (3)
Peripheral Motor Neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Mood Alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest soreness and tightness (General disorders) | 1 (1) | 0 (0)
Fungal rash (Infections and infestations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood spotting (Renal and urinary disorders) | 1 (1) | 0 (0)
Gross hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Syncopal episode with brief loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Altered taste sensation (Nervous system disorders) | 1 (1) | 0 (0)
Vein Pain (Vascular disorders) | 6 (6) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Pain, bilateral arms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain, inflammation of left arm above IV site (General disorders) | 1 (1) | 0 (0)
Aches and pains (General disorders) | 1 (1) | 0 (0)
Pain, axilla & breast (General disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 2 (2)
Sorness in upper and lower extremities (General disorders) | 1 (1) | 0 (0)
Myalgias (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Substernal chest pressure (General disorders) | 1 (1) | 0 (0)
Pain, bone and muscle (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain, abdominal (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Pain, jaw (General disorders) | 2 (2) | 0 (0)
Pain, hips and legs (General disorders) | 1 (1) | 0 (0)
Gas pains (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint pains, back and hips (General disorders) | 1 (1) | 0 (0)
Ache and heaviness in left arm (General disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Pain, right groin (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Generalized achiness (General disorders) | 2 (2) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Pain, related to PICC (General disorders) | 1 (1) | 0 (0)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain, lower back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (18) | 1 (1)
Weight loss (General disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 41 (48) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No